CLINICAL TRIAL: NCT01330654
Title: Using Heart Rate Variability to Analyze the Effect of Beta Blockers on Intermediate Risk Patients Undergoing Laparoscopic Surgical Procedures
Brief Title: Heart Rate Variability (HRV) to Evaluate Surgical Risk on Patients on Beta Blockers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patients were enrolled. Study was closed prior to study start.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Jim Davis, Interim Program Director, Department of Surgery, UCSF Fresno
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2010030
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Cardiac Event Risk
Keywords: Intermediate risk of adverse cardiac event; Undergoing laparoscopic surgical procedure; Age forty to seventy five
MeSH Terms: interventions — Metoprolol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beta blocker (Active Comparator): These patients will be randomized to receive a standard dose of metoprolol (50mg) starting two weeks prior to surgery
  Interventions: Drug: metoprolol
- Control (No Intervention): This arm will receive no additional treatment prior to surgery

INTERVENTIONS:
Drug: metoprolol — 50mg PO BID starting two weeks prior to surgery. Patients will be reevaluated one week prior to surgery. If their pulse is above 70, the dose will be increased to 100mg BID. If the HR is 50-70, the dose will not be changed. If the pulse is below 50, the dose will be decreased to 25mg. This dose will be continued for thirty days after operation.
  Arms: Beta blocker

SUMMARY:
Beta blockers have been shown to decrease the risk of intraoperative cardiac events in patients at high cardiac risk. However, they have also been associated with side effects (for instance, stroke.) The role of beta blockers in patients at intermediate cardiac risk undergoing surgery is controversial. Heart rate variability is a way of evaluating the cardiac function of a patient. Decreased heart rate variability is associated with early cardiac death in patients with congestive heart failure (CHF) and after a heart attack. It has been shown to transiently decrease in patients in hemorrhagic shock after trauma and returns to normal after resuscitation in trauma and burn patients. The investigators hypothesize that beta blockers will maintain pre operative heart rate variability in patients with intermediate risk of cardiac events during operative intervention with laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* age 40-75 years old
* intermediate risk of adverse cardiac events:

  * renal insufficiency (CrCl < 60)
  * diabetes mellitus
  * two of the following:

    * age > 50
    * obesity
    * hypertension
    * hyperlipidemia
    * hypercholesterolemia
    * prior stroke
  * undergoing an elective laparoscopic abdominal surgery less than three hours:

    * cholecystectomy
    * ventral hernia repair
    * umbilical hernia repair
    * gastric bypass or gastric banding

Exclusion Criteria:

* currently taking a beta blocker
* prior heart attack
* rhythm other than sinus on ECG
* contraindication to beta blockers:

  * decompensated CHF
  * severe valvular disease
  * asthma
  * COPD
  * hypersensitivity to beta blockers
  * heart rate < 60
* currently taking a calcium channel blocker
* urgent or emergent surgery

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Wessel, MD, Study Director — UCSF Fresno Department of Internal Medicine
Locations (1):
- Community Regional Medical Center, Fresno, California, United States

REFERENCES:
- [Background] Fleisher LA, Beckman JA, Brown KA, Calkins H, Chaikof E, Fleischmann KE, Freeman WK, Froehlich JB, Kasper EK, Kersten JR, Riegel B, Robb JF, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Hunt SA, Lytle BW, Nishimura R, Page RL, Riegel B; American College of Cardiology/American Heart Association Task Force on Practice Guidelines Writing Committee to Update the 2002 Guidelines on Perioperative Cardiovascular Evaluation for Noncardiac Surgery; American Society of Echocardiography; American Society of Nuclear Cardiology; Heart Rhythm Society; Society of Cardiovascular Anesthesiologists; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology. ACC/AHA 2006 guideline update on perioperative cardiovascular evaluation for noncardiac surgery: focused update on perioperative beta-blocker therapy: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Update the 2002 Guidelines on Perioperative Cardiovascular Evaluation for Noncardiac Surgery): developed in collaboration with the American Society of Echocardiography, American Society of Nuclear Cardiology, Heart Rhythm Society, Society of Cardiovascular Anesthesiologists, Society for Cardiovascular Angiography and Interventions, and Society for Vascular Medicine and Biology. Circulation. 2006 Jun 6;113(22):2662-74. doi: 10.1161/CIRCULATIONAHA.106.176009. No abstract available. PMID 16754815
- [Background] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210
- [Background] Kleiger RE, Miller JP, Bigger JT Jr, Moss AJ. Decreased heart rate variability and its association with increased mortality after acute myocardial infarction. Am J Cardiol. 1987 Feb 1;59(4):256-62. doi: 10.1016/0002-9149(87)90795-8. PMID 3812275
- [Background] Poldermans D, Boersma E, Bax JJ, Thomson IR, van de Ven LL, Blankensteijn JD, Baars HF, Yo TI, Trocino G, Vigna C, Roelandt JR, van Urk H. The effect of bisoprolol on perioperative mortality and myocardial infarction in high-risk patients undergoing vascular surgery. Dutch Echocardiographic Cardiac Risk Evaluation Applying Stress Echocardiography Study Group. N Engl J Med. 1999 Dec 9;341(24):1789-94. doi: 10.1056/NEJM199912093412402. PMID 10588963
- [Background] Beckers F, Verheyden B, Ramaekers D, Swynghedauw B, Aubert AE. Effects of autonomic blockade on non-linear cardiovascular variability indices in rats. Clin Exp Pharmacol Physiol. 2006 May-Jun;33(5-6):431-9. doi: 10.1111/j.1440-1681.2006.04384.x. PMID 16700875
- [Background] Yang H, Raymer K, Butler R, Parlow J, Roberts R. The effects of perioperative beta-blockade: results of the Metoprolol after Vascular Surgery (MaVS) study, a randomized controlled trial. Am Heart J. 2006 Nov;152(5):983-90. doi: 10.1016/j.ahj.2006.07.024. PMID 17070177
- [Background] POISE Study Group; Devereaux PJ, Yang H, Yusuf S, Guyatt G, Leslie K, Villar JC, Xavier D, Chrolavicius S, Greenspan L, Pogue J, Pais P, Liu L, Xu S, Malaga G, Avezum A, Chan M, Montori VM, Jacka M, Choi P. Effects of extended-release metoprolol succinate in patients undergoing non-cardiac surgery (POISE trial): a randomised controlled trial. Lancet. 2008 May 31;371(9627):1839-47. doi: 10.1016/S0140-6736(08)60601-7. Epub 2008 May 12. PMID 18479744
- See also: PhysioNet is a database of physiologic signals and contains information on heart rate variability — http://www.physionet.org